CLINICAL TRIAL: NCT03675074
Title: Single Arm Study of Neurotronic Fully Endoscopic Jejunoileal Side-to-side Anastomosis for Treatment of Obesity and Type II Diabetes: The Neujia 1A Trial
Brief Title: Neujia Anastomosis for Treatment of Obesity and Type II Diabetes
Acronym: NEUJIA 1A
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Deployment site not obtained in 5 patients with endoscopic screening and intent-to-treat. No devices implanted and no AEs through 30days.
Sponsor: Neurotronic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 450 - NEUJIA 1A Study CIP
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Type2 Diabetes Mellitus; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): A dual path jejunoileal side-to-side anastomosis is endoscopically created using the Neujia device.
  Interventions: Device: Neujia

INTERVENTIONS:
Device: Neujia — Neujia devices endoscopically deployed for jejunoileal compression anastomosis

SUMMARY:
This prospective, multicenter, open label, single arm study will enroll subjects presenting with obesity and inadequately controlled type II diabetes (T2DM). A dual path jejunoileal side-to-side anastomosis is endoscopically created using the Neujia device. Subjects are followed for 12 months and annually thereafter for up to 5 years to assess change in metabolic parameters, medications, weight, and adverse events.

DETAILED DESCRIPTION:
For many obese diabetics, medical treatment and lifestyle modification fail to provide acceptable glucose levels or durable weight loss. Bariatric surgical procedures have been proven to provide better glycemic control and to improve life expectancy and quality of life. But these are invasive procedures with significant complications, and notwithstanding the strong clinical evidence and consensus guidance, less than 2% of patients who would benefit from bariatric surgery choose to undergo the invasive procedures. There is therefore a significant unmet clinical need for metabolic/bariatric therapies that result in durable improvement in glycemic control, decreased anti-diabetic medication requirements, and weight loss, with fewer and less severe complications than invasive bariatric surgery.

Human clinical data suggests that partial diversion through a side-to-side jejunoileal anastomosis results in an absolute decrease in HbA1c of 1.9 to 3.6 percentage points and a decrease in total weight of 9.6 to 14.6% at 12 months. Although these studies used other methods, they provide good evidence that the anastomosis created by Neujia should be expected to safely improve glycemic control.

A minimally invasive anastomosis device (Neujia) and endoscopic delivery system have been developed to create a side-to-side jejunoileal anastomosis. One device is deployed in the jejunum, approximately 30 to 100 cm distal to the ligament of Treitz, and the other in the ileum, approximately 30 to 100 cm proximal to the ileocecal valve. The devices are mated under endoscopic guidance with fluoroscopic visualization and create a compression anastomosis. Neujia has the potential to provide a fully endoscopic, incisionless procedure that achieves durable weight loss and glycemic control without the risks of bariatric surgery. The proposed single arm study is designed to assess the feasibility and safety and efficacy of the Neujia device when used to treat T2DM and obesity. Subjects are followed for 12 months and annually thereafter for up to 5 years to assess change in metabolic parameters, medications, weight, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 and < 65 years, estimated life expectancy ≥ 2 years;
2. BMI ≥ 30 and < 40 kg/m2;
3. HbA1c ≥ 8.0 and ≤ 11%;
4. Fasting Glucose (FG) ≥ 126 mg/dL;
5. Under active medical care with ≥ 6-months treatment on ≥ 2 anti-diabetic medications;
6. T2DM diagnosed ≤ 10 years prior to enrollment;
7. Non-fasting random or stimulated C-peptide ≥ 2 ng/mL (660 pmol/l);
8. Willing and able to provide informed consent, comply, and be geographically stable

Major Exclusion Criteria:

1. Type I diabetes, positive autoantibodies to glutamic acid decarboxylase 65 (GAD65), secondary diabetes;
2. Hypoglycemia unawareness or serious hypoglycemia with loss of consciousness or confusion sufficient to prevent self-treatment in last 6 months;
3. Any condition for which endoscopy or colonoscopy would be contraindicated;
4. Any condition for which general anesthesia would be contraindicated;
5. Congenital or acquired anomalies of the gastrointestinal (GI) tract, abnormal GI anatomical finding, or anatomy precluding deep small bowel enteroscopy sufficient to prevent endoscopic advancement to the target treatment site;
6. Previous laparoscopic or open abdominal or pelvic surgery (except for prior caesarian section or laparoscopic cholecystectomy, which are allowed);
7. History of abdominal or pelvic infection or disease or procedures that may have resulted in abdominal adhesions;
8. Known history of autoimmune bowel disease or chronic inflammatory bowel disease (IBD);
9. Active inflammatory gastrointestinal disease (e.g., pancreatitis, hepatitis) or systemic infection (e.g., tuberculosis, malaria);
10. Known history of chronic liver disease (except nonalcoholic steatohepatitis (NASH)/ nonalcoholic fatty liver disease (NAFLD)), hepatic cirrhosis, or current transaminase/alkaline phosphatase elevation above three times the upper limit of normal (in the absence of NASH/NAFLD);
11. Severe or unstable pulmonary or circulatory comorbidities posing risks to the patient that may confound the results of the study in investigator's judgment;
12. History of cardiovascular event within last 6 months or with chronic sequela;
13. Uncontrolled hypertension with systolic blood pressure (SBP) over 160 mmHg or diastolic blood pressure (DBP) over 110 mmHg;
14. Estimated glomerular filtration rate (eGFR) < 30 mL/min per 1.73 m2;
15. Currently taking pre-meal, bolus, or premixed insulin (patients on basal insulin only are allowed);
16. Malignancy that required therapy in the last 5 years (unless cancer only in situ e.g. basal cell carcinoma (BCC)), history of organ transplantation, or currently on immune-suppressive, chemotherapeutic, or radiation therapy;
17. History of vasculopathy, coagulopathy, or currently on anti-coagulation therapy;
18. Abnormal wound healing, e.g., human immunodeficiency virus (HIV), corticosteroid, or immunosuppressive agent use;
19. Planned magnetic resonance imaging (MRI) or any condition for which MRI is likely to be indicated within 3 months;
20. Pregnant or planning on becoming pregnant within 12 months of procedure;\
21. Known serious or uncontrolled psychiatric disease, eating disorder, or active alcohol or drug addiction.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months

SECONDARY OUTCOMES:
Technical and Procedural Success | 1 day
  Successful endoscopic deployment without procedural serious adverse events
Composite Safety: percent of subjects with Freedom from bowel perforation, anastomotic leak, stricture, obstruction, and prolonged dumping syndrome (>90 days) | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
Reversal or Revision Rate | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
Change in HbA1c | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
Change in diabetic medications | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
  Change in the number of prescribed anti-diabetic medications and dosage from subject's medications at baseline
Percentage with HbA1c ≤ 6.5% or ≤ 7.0%, by medication status | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
Change in fasting plasma glucose (FG) | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
Change in weight | 1, 3, 6, 9, 12, 24, 36, 48, 60 months

OTHER OUTCOMES:
Improvement in metabolic comorbidities | 1, 3, 6, 9, 12, 24, 36, 48, 60 months
  Change in severity and required medications to treat metabolic comorbidities such as hypertension, dyslipidemia, etc...

CONTACTS AND LOCATIONS:
Overall Officials: Irving Waxman, MD, Principal Investigator — Center Director of The Center for Endoscopic Research and Therapeutics (CERT), University of Chicago Medicine